CLINICAL TRIAL: NCT05987631
Title: Preoperative Predictors of Weight Loss and Improved Metabolic Health After Bariatric Surgery
Brief Title: Predictors of Weight Loss and Metabolic Health After Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Obesitas Kliniek B.V. (Unknown); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Mireille JM Serlie, Prof. Dr. Mireille JM Serlie, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2021_136; NL77692.018.21 (Other: Amsterdam UMC); NTR9447 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2023-04-21; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Obesity, Morbid; Insulin Sensitivity; Bariatric Surgery Candidate; Feeding Behavior
Keywords: Obesity; Bariatric Surgery; Metabolic health; Weight loss; Predictors
MeSH Terms: conditions — Obesity, Morbid; Insulin Resistance; Feeding Behavior; Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and tissue (fat, muscle, liver)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study the investigators aim to identify preoperative predictors of improvement of metabolic health and weight loss after bariatric surgery focusing on inflammation, insulin sensitivity (in a subgroup of patients), glucoregulatory determinants, psychological traits, feeding behavior characteristics and cardiorespiratory fitness

DETAILED DESCRIPTION:
Obesity is the result of a complex interplay between genetic and epigenetic predisposition, environment, physical activity, nutrition and psychology. It is a debilitating disorder and a risk factor for the development of metabolic disorders such as dyslipidaemia, hypertension and hyperglycaemia as well as certain cancers. Bariatric surgery has proven to be the most effective treatment for morbid obesity with established long-term results of weight loss, remission of comorbid conditions and the improvement of Quality of Life (QoL). However, variability in these results after bariatric surgery is well known. Identifying preoperative predictors of postoperative weight loss and metabolic health is of clinical priority. Predictors could help further improve the efficacy of care for obesity by tailoring treatment to the individual, based on their predicted response and therefore optimize outcome after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Patient is ≥ 18 and ≤ 75 years old
* BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with obesity related comorbidity
* Scheduled for primary bariatric procedure: Roux-en-Y gastric bypass (RYGB) or Sleeve Gastrectomy (SG)
* Stable weight 3 months prior to inclusion weight (<10% change in body weight for 3 months prior to assessments)

In order to be eligible to participate in the subgroup of this study, we will use the following inclusion criteria:

* Ability to provide informed consent
* Patient is ≥ 18 and ≤ 75 years old
* BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 with obesity related comorbidity
* Patients scheduled for RYGB
* Patients who are insulin resistant (impaired fasting glucose (> 5.6 mmol/L) or fasting insulin > 74 pmol/L)
* Postmenopausal women (to prevent bias due to the effect of sex hormones on insulin sensitivity)

Exclusion Criteria:

* Any actual medical condition except for obesity related health issues or well treated hypothyroidism
* Pregnancy anticipated in the first two years following surgery

A potential subject who meet the following criteria will be excluded from participation in the subgroup of this study:

* Coagulation disorders and/or use anticoagulants
* Use of any medication except for statins, antihypertensives (except for Angiotensine converting enzyme (ACE)- or angiotensin receptor blockers) and thyroid hormone
* Diabetes mellitus type 2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Nederlandse Obesitas Kliniek (Dutch Obesity Clinic).
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Predictors of improvement in metabolic health - insulin sensitivity | Baseline up to 5 years after surgery
  HOMA-IR
Predictors of improvement in metabolic health - level of glucose control | Baseline up to 5 years after surgery
  HbA1C (mmol/mol)
Predictors of improvement in metabolic health - glucose | Baseline up to 5 years after surgery
  Fasting glucose (mmol/L)
Predictors of improvement in metabolic health - insulin | Baseline up to 5 years after surgery
  Insulin (pmol/L)
Predictors of improvement in metabolic health - lipid profile | Baseline up to 5 years after surgery
  Lipids (mmol/L)
Predictors of improvement in metabolic health - biomarker inflammation | Baseline up to 5 years after surgery
  CRP (mg/L)
Predictors of improvement in metabolic health | Baseline up to 5 years after surgery
  Genetic variants using GWAS analysis
Predictors of weight loss | Baseline up to 5 years after surgery
  Genetic variants using GWAS analysis

SECONDARY OUTCOMES:
Psychological factors - depression | Baseline up to 5 years after surgery
  Patient-Reported Outcomes Measurement Information System Depression (PROMIS-D: validated questionnaire for bariatric surgery. PROMIS-D: range in score from 8 to 40, higher scores indicating greater severity of depression
Psychological factors - anxiety | Baseline up to 5 years after surgery
  Patient-Reported Outcomes Measurement Information System Anxiety (PROMIS-A): validated questionnaire for bariatric surgery. PROMIS-A: range in score from 7 to 35, higher scores indicating greater severity of anxiety.
Psychological factors - impulsivity | Baseline up to 5 years after surgery
  Measurements of impulsiveness Barret Impulsiveness Scale (BIS): validated questionnaire to assess level of impulsivity
  BIS-11: The total scores can range from 30 to 120. Higher scores on the BIS reflect higher levels of impulsiveness.
Psychological factors - impulsivity | Baseline up to 5 years after surgery
  Measurements of impulsiveness Iowa Gambling Task: validated task to study impulsive behaviour
  Iowa gambling task: The net score is calculated by subtracting the number of disadvantageous selections from the advantageous selections. A positive net score indicates better performance
Predictors of weight loss - food addiction | Baseline up to 5 years after surgery
  Food addiction scale (YFAS 2.0): validated questionnaire to assess food addiction.
  YFAS 2.0 includes two scoring methods, a continuous symptom count and a diagnosis of food addiction.
  Continious symptom count ranges from zero to eleven, Diagnosis of food addiction: no food addiction (0-1 symptoms), a mild food addicition (2-3 symptoms), a moderate food addiction (4-5 symptoms), or a severe food addiction (>6 symptoms).
Predictors of weight loss - eating behaviour | Baseline up to 5 years after surgery
  Dutch Eating Behaviour Questionnaire (DEBQ): validated questionnaire to assess eating behaviour.
  DEBQ consists of 33 items.Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
Predictors of weight loss - Quality of Life | Baseline up to 5 years after surgery
  Selfesteem scale of Impact of Weight on Quality of Life - lite (IWQOL-lite): validated questionnaire after weight loss interventions. The self-esteem scale consists of 7 items. Each item is rated on a 5-point scale. Higher scores represent better quality of life.
Predictors of weight loss - Quality of Life | Baseline up to 5 years after surgery
  OBESI-Q (Obesity): validated questionnaire for reporting Health Related Quality of Life. Outcome is expressed on a 100 point scale, a higher score is higher quality of life, with the exception of item "Excess skin".
Predictors of weight loss - Quality of Life | Baseline up to 5 years after surgery
  EuroQuality of Life (EQ-5D): validated questionnaire for reporting Quality of Life after bariatric surgery. Each item is rated on a 5-point scale. Higher scores represent lower reported quality of life.
Predictors of weight loss - Impulsivity | Baseline up to 5 years after surgery
  Measurements of impulsiveness Barret Impulsiveness Scale (BIS): validated questionnaire to assess level of impulsivity
  BIS-11: The total scores can range from 30 to 120. Higher scores on the BIS reflect higher levels of impulsiveness.
Predictors of weight loss - Impulsivity | Baseline up to 5 years after surgery
  Measurements of impulsiveness Iowa Gambling Task: validated task to study impulsive behaviour
  Iowa gambling task: The net score is calculated by subtracting the number of disadvantageous selections from the advantageous selections. A positive net score indicates better performance
Predictors of weight loss - Physical activity | Baseline up to 5 years after surgery
  Short Questionnaire to Assess Health Enhancing Physical Activity (SQUASH): validated questionnaire to assess physical activity.
  The SQUASH measures the frequency, duration and intensity of 5 different physical activities: commuting (traveling to and from work/study), housekeeping , activities at work, leisure time, and sports. A higher score = more time spend on physical activities.
Sexual dimorphism in weight loss | Baseline up to 5 years after surgery
  Males versus females regarding weight loss (kg) and percentage of total weight loss
Sexual dimorphism in restoration of metabolic health - insulin sensitivity | Baseline up to 5 years after surgery
  Males versus females regarding insulin sensitivity (HOMA-IR) and measurements of glucose and insuline
Sexual dimorphism in restoration of metabolic health - improvement of diabetes | Baseline up to 5 years after surgery
  Males versus females regarding HbA1c values and diabetic drug use
Sexual dimorphism in restoration of metabolic health - lipid | Baseline up to 5 years after surgery
  Males versus females regarding lipids (mmol/L) and lipid-lowering agents use
Sexual dimorphism in restoration of metabolic health - hypertension | Baseline up to 5 years after surgery
  Males versus females regarding blood pressure (mmHg) and anithypertensive medication use
Peripheral insulin sensitivity | Before and 3 and 18 months after bariatric surgery
  In a subset of 40 patients insulin sensitivity will be assessed using hyperinsulinemic euglycemic clamps, and adipose tissue and skeletal muscle biopsies will be taken to assess insulin signalling (expression of mRNA and phosphorylated proteins)

CONTACTS AND LOCATIONS:
Overall Officials: Mireille JM Serlie, Prof. Dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Valerie M Monpellier, Dr., Principal Investigator — Obesitas Nederland B.V.
Locations (3):
- Netherlands (3):
  - Nederlandse Obesitas Kliniek Gouda, Gouda, South Holland
  - Nederlandse Obesitas Kliniek Den Haag, The Hague, South Holland
  - Nederlandse Obesitas Kliniek Nieuwegein, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided